CLINICAL TRIAL: NCT03327623
Title: A Prevalence and Incidence Study Investigating the Burden of Atrial and Ventricular Arrhythmias in Patients With Hypertrophic Cardiomyopathy and Sleep Apnea.
Brief Title: Sleep Apnea and Hypertrophic Cardiomyopathy (HCM)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Principal Investigator, Mayo Clinic
Other Study IDs: 17-003514; 1R01HL134885-01 (NIH)
Record Dates: First submitted 2017-10-25; First posted 2017-10-31 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: sleep apnea; arrhythmia
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Sleep Apnea Syndromes; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma, serum and urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertrophic Cardiomyopathy (HCM): Subjects with a diagnosis of Hypertrophic Cardiomyopathy
- Control: Subjects who are healthy volunteers

SUMMARY:
The investigators are trying to find out how common sleep apnea is in hypertrophic cardiomyopathy. The purpose of this study is to see if sleep apnea is common in hypertrophic cardiomyopathy and if its presence is associated with changes in the functioning of the body. The investigators want to determine if sleep apnea is associated with electrical disorders of the heart in patients with hypertrophic cardiomyopathy.

DETAILED DESCRIPTION:
Participants will be healthy volunteers or subjects with the diagnosis of hypertrophic cardiomyopathy (HCM). All patients will a undergo a one time; medical history, physical examination, questionnaires, sleep observation in hospital, blood and urine samples, ultrasound scan of the heart, paced breathing test, ultrasound of brachial artery in the arm, MRI of the heart & 48 hour ECG Holter monitoring. Comparison between the normal volunteers and subjects with HCM will be made.

ELIGIBILITY:
Inclusion criteria:

* Adults with a diagnosis of HCM
* Able to consent
* Non-pregnant
* Healthy Controls free of hypertrophic cardiomyopathy and without a definitive family history of hypertrophic cardiomyopathy.

Exclusion criteria:

* Decompensated Heart failure at time of enrollment (prior history of HF is not an exclusion criteria)
* Severe (known) Chronic obstructive pulmonary disease (COPD) (FEV1 between 30 and 50 percent of normal)
* Vulnerable study populations except for minorities (minorities may be targeted to achieve 25% minority recruitment required by the NIH)
* Pregnant women
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and Subjects from The Mayo Clinic Hypertrophic Cardiomyopathy (HCM) Registry who reside in Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Prevalence of Obstructive Sleep Apnea (OSA). | Approximately 2 years.
  Measured by the Apnea-hypopnea index (AHI). The AHI is the number of apneas or hypopneas recorded during the study per hour of sleep. It is generally expressed as the number of events per hour. Based on the AHI, sleep apnea is diagnosed if an AHI ≥5 events/hour.
Determine the severity of Sleep Apnea. | Approximately 2 years.
  The severity of OSA is classified based on the AHI as follows: None/Minimal: AHI < 5 per hour, Mild: AHI ≥ 5, but < 15 per hour, Moderate: AHI ≥ 15, but < 30 per hour, Severe: AHI ≥ 30 per hour.
Differences in Autonomic Regulation. | Approximately 2 years.
  In persons with hypertrophic cardiomyopathy and sleep apnea vs. those without sleep apnea.
Prevalence of atrial arrhythmias. | Approximately 2 years.
  Investigators will determine prevalence of atrial arrhythmias, based on prior ECG documented atrial arrhythmias at any timepoint prior to enrolment and up to 4 weeks after the study date. Participants will also have a 48h ECG (extended Holter) recorder attached to screen for atrial arrhythmias.
Incidence of atrial arrhythmias. | Approximately 5 years.
Frequency of ventricular arrhythmias. | Approximately 5 years.
  Investigators will prospectively follow patients with hypertrophic cardiomyopathy to determine the frequency of ventricular arrhythmias in those with vs those without sleep apnea.

SECONDARY OUTCOMES:
Identify novel biomarkers | Approximately 5 years
  Participants will be prospectively followed and blood collected to identify biomarkers of arrhythmia, heart failure and prognosis in persons with hypertrophic cardiomyopathy.
Investigate the association of sleep apnea with atrial and ventricular fibrosis | Approximately 7 years
  Participants will undergo baseline MRI studies of the heart to determine the burden of fibrosis and its association with sleep apnea. Participants may be invited to complete a follow-up study to track changes in fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No